CLINICAL TRIAL: NCT04037475
Title: Treatment of Herpes Labialis by Photodynamic Therapy: Controlled, Prospective, Randomized, Double-blind Protocol Study
Brief Title: Treatment of Herpes Labialis by Photodynamic Therapy
Acronym: Herpes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Anna Carolina Ratto Tempestini Horliana, PhD, Postgraduate program professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Herpes
Record Dates: First submitted 2019-07-24; First posted 2019-07-30 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Photodynamic Therapy; Herpes Simplex, Labial
Keywords: photodynamic therapy; herpes labialis; herpes simplex; laser
MeSH Terms: conditions — Herpes Labialis; Herpes Simplex

STUDY DESIGN:
Intervention Model Description: 24 individuals will be randomly divided into 2 groups: G1 (control group) - conventional treatment with acyclovir and simulation of treatment with photodynamic therapy; G2 (experimental group) - photodynamic therapy placebo ointment simulating acyclovir cream.
Who Masked: Participant, Investigator
Masking Description: Only the researcher responsible for performing the treatments (which will open the envelopes of the randomization) will know which treatment was assigned to each patient. The identification of each group will be revealed only after the statistical analysis of the data for all those involved in the study by this researcher. Therefore, the researcher responsible for data collection, the microbiologist and the statistician will be blind regarding the treatments assigned to the groups. The patient will also be blind to the type of treatment performed, since the treatment of the lesion will be identical in both groups and the treatment with PDT will be simulated in the control group. Aciclovir placebo will be used in the experimental group, so the patient will not know which treatment will be effective.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (placebo) (Placebo Comparator): The patients will receive an agent with the same vehicle as methylene blue to mimic irrigation with the photosensitizer and the laser will be switched off at the time of application. The placebo PDT procedures will be performed on the lesion: Application of methylene blue placebo with a carpule syringe and needle (with stop and without bevel) inside the lesions; 1 minute of pre-irradiation will be expected. The irradiations will be performed with the same device positioned in the same way and at the same time of application, however, the laser will be turned off. The beep sound will be recorded and turned on during application to blind treatment to the patient. The patient will receive a catheter with acyclovir cream and will be advised to spread on the lesions four times a day for 7 days, which will be their return for reevaluation. It will be washed in abundance with saline (saline solution) until the total removal of the placebo from the photosensitizer.
  Interventions: Device: photodynamic therapy herpes labialis
- experimental group (Experimental): Patients will be treated with photodynamic therapy and will receive a placebo ointment simulating acyclovir cream. If the lesions are in the vesicle phase, they will be ruptured with a sterile needle. The methylene blue solution at 0.005% concentration will be gently placed on the lesions. Application of methylene blue on the lesions.1 minute of pre-irradiation will be expected. The irradiations will be performed with the Laser Duo® with a wavelength of 660 nm, with a power of 100 mW(milliwatts), the energy density of 300 J / cm², with the energy of 3 J (joules) in the center of the lesion for 30 seconds. The laser will be positioned in direct contact with the lesion, perpendicular, applied centrally to each lesion with energy per point of 3J. Wash in abundance with saline solution until the removal of the photosensitizer is complete. Patients will receive a tube with a placebo cream simulating aciclovir and the same will be advised to spread the cream 4 times per day for 7 days.
  Interventions: Device: photodynamic therapy herpes labialis

INTERVENTIONS:
Device: photodynamic therapy herpes labialis — Patients will receive Photodynamic Therapy (PDT), irradiations will be performed with the Laser Duo® red laser diode (MMOptics, São Carlos, SP, Brazil) with a wavelength of 660 nm, with a power of 100 mW, the energy density of 300 J / cm², with energy of 3 J in the center of the lesion for 30 seconds. The laser will be positioned in direct contact with the lesion, perpendicular, applied centrally to each isolated lesion that presents with fixed energy per point of 3J. Wash in abundance with saline solution until the removal of the photosensitizer is complete. All treatment proposed in group 1 (simulation of PDT + delivery of aciclovir cream) in each patient will be concluded in a single session. Treatment for group 2 (PDT + placebo cream) will also be completed in a single session. All possible adverse effects will be noted and qualified during the treatment protocol and maintenance period (3/3 months) using the questionnaire developed for this protocol.

SUMMARY:
Lesions of herpes labialis are caused by the herpes simplex virus type 1 (HSV-1) and cause pain and aesthetic compromise. It is characterized by the formation of small vesicles that coalesce and rupture forming extremely painful ulcers, that evolve to crusts, dry desquamations until their complete remission. Currently, the treatment of these lesions is done with acyclovir. Although it diminishes the symptomatology, it causes viral resistance and does not prevent the recurrence of the lesions. It is known that photodynamic therapy (PDT) has numerous advantages, among them: the reduction of the time of remission, and does not cause resistance.

A total of 30 patients with herpes labialis in the prodromal stage of vesicles, ulcers, and crusts will be selected to participate in the study and randomized into two groups: G1 control and G2 experimental. After signing informed consent, patients in group G1 will undergo the standard gold treatment for cold sores with acyclovir and simulated PDT treatment. Patients in the experimental G2 group will be treated simulating the gold standard treatment of herpes labialis (placebo) and PDT.

DETAILED DESCRIPTION:
Lesions of herpes labialis are caused by the herpes simplex virus type 1 (HSV-1) and cause pain and aesthetic compromise. It is characterized by the formation of small vesicles that coalesce and rupture forming extremely painful ulcers, that evolve to crusts, dry desquamations until their complete remission. Currently, the treatment of these lesions is done with acyclovir. Although it diminishes the symptomatology, it causes viral resistance and does not prevent the recurrence of the lesions. It is known that photodynamic therapy (PDT) has numerous advantages, among them: the reduction of the time of remission, and does not cause resistance.

Materials and methods: A total of 30 patients with herpes labialis in the prodromal stage of vesicles, ulcers, and crusts will be selected to participate in the study and randomized into two groups: G1 control and G2 experimental. After signing TCLE and TA, patients in group G1 will undergo the standard gold treatment for cold sores with acyclovir and simulated PDT treatment. Patients in the experimental G2 group will be treated simulating the gold standard treatment of herpes labialis (placebo) and PDT. In all patients will be collected saliva samples for analysis of cytokines, and will be performed exfoliative cytology in the lesions. The pain will be assessed through a pain scale and a questionnaire of quality of life-related to oral health (Ohip- 14) will be given to them. Patients will continue to be followed up after 7 days, 1 month, 3 months, 6 months and 1 year and, if there is a recurrence of the lesion, they will contact the researchers.

ELIGIBILITY:
Inclusion Criteria:

- Patients of both sex,

* with no predilection for race or socioeconomic status,
* negative medical history

Exclusion Criteria:

* Patients with a herpes infection in the dry desquamation stage will be excluded.
* Participants in continuous use of non-steroidal anti-inflammatory drugs and continued corticosteroid therapy for less than 1 week.
* Diabetic participants, smokers
* who need immunosuppressants,
* pregnant women and/or nursing mothers.
* HIV positive,
* hepatitis B or C.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of the resolution time of the lesions | through study completion on average of one year
  Evaluation of the resolution time of the lesions in days (primary objective of the study). For this, a 15-day follow-up will be performed for this variable.The complete resolution will be accompanied by photos and telephone contact and noted in a specific clinical file. For this, a 1-year follow-up will be performed for this variable. The location of the lesions through sextants on the lips (sextants 1, 2 and 3 to upper left to right and sextants 4,5 and 6 from right to left, with sextant 2 in the labial filter region and sextant 5 is its lower lip antagonist.

SECONDARY OUTCOMES:
Evaluate if the amount of HSV-1 decreases after treatment with PDT | through study completion on average of three years
  by qPCR (polymerase reaction ) at the baseline (T0), 3 (T1) and 7 (T2).HSV lesion secretion samples will be collected at 1 single site in the central portion of the lesion with sterile swab after treatment of all HSV lesions. They will be stored in 500 μl of Tris-EDTA (ethylenediamine tetraacetic acid) in tubes of 1 , 5ml for microcentrifuge (Eppendorff®). During the collection period (in the clinic) the samples will be stored on ice inside a styrofoam. These samples will be properly identified and stored at -80ºC (centigrades) (freezer from the UNINOVE University nove de Julho Biophotonics Laboratory) until further analysis.
evaluation of saliva cytokines IL-6, IL-1β, IL-8, TNF-α (tumor necrosis factor) and IL-10 (interleukine) | through study completion on average of three years
  by ELISA method in non-stimulated saliva in the baseline (T0), 3 (T1) and 7 T2) and 30 days after treatment (T3).Samples of unstimulated saliva (2 ml) will be collected in 50 ml tubes (Falcon tube). In the laboratory 500 μl of pure saliva will be added to 500 μl TE (tris-EDTA), and stored at -80 ° C (freezer from the UNINOVE Biophotonics laboratory).
presence of pain: visual analog scale | through study completion on average of three years
  verify the pain by visual analog scale at baseline (T0), 3 (T1) and 7 (T2) and 30 days after treatment (T3).Will be assessed by applying the visual analogue scale (EVA) with a line of 100 mm, with both ends closed. One end has the indication "0" and the other "10" which means respectively no pain and unbearable pain. Instructions for marking will always be given to the patient by the same operator. Each patient will be instructed to mark with a vertical trace the point that best corresponds to the intensity of pain at the time of evaluation
Oral health impact profile (Ohip-14) | through study completion on average of three years
  This questionnaire is a simplified form of the original OHIP-49 questionnaire, the Ohip-14, and will be used to assess the impact of oral health on the quality of life of the research participants. The Ohip-14 is used to measure perceived needs. It measures the impact of oral changes on oral health related quality of life. The patient responds to 14 questions by assigning to his answers the values 0 (never), 1 (almost never), 2 (sometimes), 3 (most of the time) and 4 (always)
Temperature | through study completion on average of three years
  The temperature will be measured at the site of the lesion (at its central point) and at its side (healthy skin 2 cm from the edge of the lesion). The local measurement will be measured using the Safety 1st® digital thermometer (Safety 1st®, "No Touch Forehead", Columbus, USA
evaluation of HSL lesions cytokines IL-6, IL-1β, IL-8, TNF-α (tumor necrosis factor) and IL-10 (interleukine) | through study completion on average of three years
  by ELISA method in HSL lesions in the baseline (T0), 3 (T1) and 7 T2) and 30 days after treatment (T3).Samples of unstimulated saliva (2 ml) will be collected in 50 ml tubes (Falcon tube). In the laboratory 500 μl of pure saliva will be added to 500 μl TE (tris-EDTA), and stored at -80 ° C (freezer from the UNINOVE Biophotonics laboratory).

CONTACTS AND LOCATIONS:
Locations (1):
- Anna Carolina R.T. Horliana, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ramalho KM, Rocha RG, Correa-Aranha AC, Cunha SR, Simoes A, Campos L, Eduardo Cde P. Treatment of herpes simplex labialis in macule and vesicle phases with photodynamic therapy. Report of two cases. Photodiagnosis Photodyn Ther. 2015 Jun;12(2):321-3. doi: 10.1016/j.pdpdt.2015.02.005. Epub 2015 Mar 10. No abstract available. PMID 25770054
- [Result] Marotti J, Aranha AC, Eduardo Cde P, Ribeiro MS. Photodynamic therapy can be effective as a treatment for herpes simplex labialis. Photomed Laser Surg. 2009 Apr;27(2):357-63. doi: 10.1089/pho.2008.2268. PMID 19382840
- [Result] Palmieri M, Ornaghi M, Martins VAO, Correa L, Brandao TB, Ribeiro ACDP, Sumita LM, Tozetto-Mendoza TR, Pannuti CS, Braz-Silva PH. Oral shedding of human herpesviruses in patients undergoing radiotherapy/chemotherapy for head and neck squamous cell carcinoma is not affected by xerostomia. J Oral Microbiol. 2018 May 28;10(1):1476643. doi: 10.1080/20002297.2018.1476643. eCollection 2018. PMID 29868164
- [Derived] La Selva A, Bezerra DT, Zerbinati RM, Goncalves MLL, Navarro RS, Bello-Silva MS, Ando-Suguimoto ES, Aranha ACC, Braz-Silva PH, Ramalho KM, Motta LJ, Fernandes KPS, Bussadori SK, Mesquita-Ferrari RA, Frochot C, Horliana ACRT. Herpes Simplex Treated With Antimicrobial Photodynamic Therapy: Randomized Controlled Trial. J Oral Pathol Med. 2025 Aug;54(7):547-555. doi: 10.1111/jop.13647. Epub 2025 Jun 8. PMID 40485092
- [Derived] La Selva A, Negreiros RM, Bezerra DT, Rosa EP, Pavesi VCS, Navarro RS, Bello-Silva MS, Ramalho KM, Aranha ACC, Braz-Silva PH, Fernandes KPS, Bussadori SK, Horliana ACRT. Treatment of herpes labialis by photodynamic therapy: Study protocol clinical trial (SPIRIT compliant). Medicine (Baltimore). 2020 Mar;99(12):e19500. doi: 10.1097/MD.0000000000019500. PMID 32195950